CLINICAL TRIAL: NCT04133090
Title: Comparison of Treatment Outcomes of Autogenous Block Bone Graft and Screw Tent-Pole Technique in Combination With Injectable Platelet Rich-Fibrin on Posterior Atrophic Mandible: A Split-Mouth Randomized Study
Brief Title: Comparison of Autogenous Bone Graft and Screw Tent-Pole Technique on Atrophic Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dentistry
Record Dates: First submitted 2019-10-16; First posted 2019-10-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Alveolar Bone Loss
Keywords: Bone augmentation; Autogenous block bone graft; Leukocytes and platelet-rich fibrin; Injectable platelet rich fibrin; Tent-pole technique
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: Split-mouth study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous block bone graft (Active Comparator): Surgical site as control group was treated with autogenous block bone graft. Augmentation site was covered with a mixture of particulate allograft and leukocyte and platelet-rich fibrin (L-PRF) membrane.
  Interventions: Procedure: Autogenous block bone graft
- i-PRF enriched allograft material+screw tent pole technique (Active Comparator): Surgical site as test group was treated with injectable platelet rich-fibrin (i-PRF) enriched allograft material. To avoid soft tissue collapse, screws were used. Augmentation site was covered with leukocyte and platelet-rich fibrin (L-PRF) membrane.
  Interventions: Procedure: i-PRF enriched allograft material+ screw tent pole technique

INTERVENTIONS:
Procedure: Autogenous block bone graft — Vertical and horizontal osteotomies were performed by means of a 6-mm diameter separation disc under copious irrigation with saline.The harvested bone graft was immediately placed in sterile saline solution to prevent dehydration. Sharp edges around the block graft were rounded under saline irrigation using a 4-mm round bur. The screw holes were properly made on both the recipient site and the block graft using a 1.3 mm drill. The graft was firmly fixed with 1.3 mm screws and a compatible driver. The periphery of the graft and the underlying gap between the screws and the recipient site, were covered with a mixture of particulate allograft and sterile saline solution to minimize resorption and to improve the adaption of the graft. All augmentation sites were covered by L-PRF membrane and flap closure was effected with 4/0 silk suture.
  Arms: Autogenous block bone graft
Procedure: i-PRF enriched allograft material+ screw tent pole technique — The i-PRF preparation was performed as follows: the blood sample collected in an 8 ml, non-coated plastic tube without anticoagulant was immediately centrifuged at a protocol of 2700 rpm for 2 min. After centrifugation, the liquid autologous fibrin material which comprised the 1 mL upper layer of the tube was collected, using a disposable syringe. The screw holes were made on the recipient site using a 1.3 mm drill. 7 mm long screws were fixed 2mm or 4mm higher than on the recipient site to provide the desired augmentation distance and stabilized by a compatible driver. i-PRF was mixed with allograft material in a sterile metal box. Polymerization was done in 3 to 5 minutes, then this material was applied to the underlying gap between the screws and the recipient site.All augmentation sites were covered by L-PRF membrane and flap closure was effected with 4/0 silk suture.
  Arms: i-PRF enriched allograft material+screw tent pole technique

SUMMARY:
The purpose of the present study was to assess the effect of injectable platelet-rich fibrin (i-PRF) enriched with allograft on alveolar bone regeneration when compared with autogenous block bone graft, in the same participants.

The study was designed as a split-mouth randomized controlled trial. The patients were randomly assigned to one of two surgical groups: the test group with i-PRF enriched particulate allograft using the screw tent-pole technique; and the control group with autogenous block bone harvested from the ramus area. All augmentation sites covered by leukocytes-PRF (L-PRF) membrane. The primary outcome variable of this study was the radiographic and histologic data collected at postoperative 6 months. The secondary outcome variable was nerve alterations and implant survival.

DETAILED DESCRIPTION:
Alveolar bone loss which results from tooth extraction, trauma or age-related factors, gives rise to the functional or structural inefficiency of implant-supported prosthetic rehabilitation. Therefore, bone augmentation techniques and graft materials are required to improve esthetic outcomes and long-term prognosis of dental implant treatment. The purpose of the present study is to evaluate the effect of i-PRF enriched with allograft on bone regeneration when compared with autogenous block bone graft. The hypothesis of the study is that i-PRF enriched with allograft will provide similar results to autogenous block bone graft for three dimensional bone reconstruction. This split-mouth randomized study was conducted in the Department of Oral Surgery of the School of Dentistry. The research protocol and informed consent forms for all procedures on patients, were approved by the local ethics committee of the University in accordance with the Helsinki Declarations of 1983.Selection of the participants was determined by clinical and radiological examination according to the inclusion criteria.Before augmentation surgery, the treatment allocation of bilateral posterior atrophic mandibles were randomly assigned to one or other of the two surgical sides: either the test group ( i-PRF + particulate allograft with screw tent-pole technique + L-PRF) or the control group (autogenous block bone graft + L-PRF) by use of the computer-generated method. Blood samples from thirteen participants were collected by a nurse at the beginning of the surgery.The L-PRF preparation was performed as follows; the venous blood samples were collected in 9 ml x 4 glass tubes without anticoagulant and immediately centrifuged at 2700 rpm for 12 min. After the centrifugation of the samples, the red blood cells (RBC) and platelet-poor plasma (PRP) were separated from the 'buffy coat' described as L-PRF. Then the L-PRF was placed on a special press kit to obtain membrane form.

Non-coated, 8 ml plastic tube without anticoagulant was immediately centrifuged at 2700 rpm for 2 min to obtain i-PRF. Following centrifugation, i-PRF was collected the tube by using a disposable syringe and mixed with allograft material. All surgeries were performed under local anesthesia. A mid-crestal incision was made on either side to expose the edentulous alveolar ridge. Furthermore, a posterior releasing incision was made over the external oblique ridge to provide access to the donor site, in control group.

Control site was treated with autogenous block bone graft and the opposite side (test site) was treated with I-PRF enriched allograft material. L-PRF membrane was used to cover augmentation sites.

The primary outcome variables of this study were the radiographic changes of augmented bone at postoperative 6 months as well as the percentage of newly formed bone, graft material and residual bone in the groups.

The secondary outcome variables were the clinical data on implant survival rate and nerve alterations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who refused to use a partially removable prosthesis and requested dental implant treatment,
* Patients had bilateral, moderate or severe posterior atrophic mandible,
* Patients had precluded conditions suitable for short dental implant.

Exclusion Criteria:

* Patients who had systemic diseases (osteoporosis, hemophilia, anemia, etc.),
* Patients who required drugs (bisphosphonate or steroid therapy),
* Patients who had a smoking habit,
* Patients who had received radiation therapy within the last two years,
* Patients who were under 18 years old, pregnant or lactating,
* Patients who had a total platelet count lower than 150,000/mm3.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
Assessment of radiological changes | Change of alveolar bone height at 6 months
  Radiologic analysis was performed to compare the changes in height of alveolar bone between the study groups
Histological assessment | Postoperatively 6 months
  Bone core samples were harvested from the implant placement sites for calculate the relative quantification of newly-formed bone within both groups as a percentage

SECONDARY OUTCOMES:
Clinical assessment | 6 months, 12 months
  Implant survival
Clinical assessment | 1 month, 6 months, 12 months
  Incidence of nerve damage were analyzed by six different sensory tests carried out three times for each evaluation area on the chin

IPD SHARING:
Plan to Share IPD: No